CLINICAL TRIAL: NCT03786016
Title: Evaluating Risk Factors and Biomarkers for Adaptation and Resilience to Spaceflight: Emotional Valence and Social Processes in Isolated, Confined and Controlled Environments
Brief Title: Evaluating Risk Factors and Biomarkers for Adaptation and Resilience to Spaceflight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Pittsburgh (Other); National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NASA80NSSC17K0644
Record Dates: First submitted 2018-12-14; First posted 2018-12-24 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Resilience; Mood; Performance; Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: All participants will be exposed to the same condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8-Days in an Isolation, Confinement Unit (Experimental): Subjects will spend 7-night/8-day in an isolated and confined unit with up to 3 other subjects.
  Interventions: Behavioral: 8-Days in an Isolation, Confinement Unit

INTERVENTIONS:
Behavioral: 8-Days in an Isolation, Confinement Unit — Subjects will spend 8 days/7 nights continuously in an isolated and confined unit with up to 3 other subjects. Subjects will participate in daily, timed activities such as space-relevant computer simulations, team tasks, and cognitive performance testing. Subjects will also experience altered environmental conditions (such as changes in lighting, sound and ambient temperature) while in the isolation unit. Subjects will receive orders from "mission control" who will monitor activity in the isolation unit and direct subjects throughout the 8-day study.

SUMMARY:
This study assesses differences in biological and behavioral domains that relate to individual adaptation and resiliency to an isolated, confined and controlled environment, and evaluates the effect of confinement, work, monotony, and social and physical isolation on stress resiliency and well-being.

DETAILED DESCRIPTION:
The goal of this study is to obtain novel information that will be used to help identify individuals who are resilient to the stressors of prolonged human spaceflight, thereby encouraging the successful completion of exploration missions and the preservation of health over the life of an astronaut. This study leverages the National Institute of Mental Health (NIMH) Research Domain Criteria (RDoC) heuristic framework to conduct experimental studies to identify biological domains (molecular, circuitry, physiology) and behavioral domains that relate to individual adaptation and resiliency (as well as behavioral vulnerability) in spaceflight-relevant confined environments. This study focuses specifically on differences among participants in their tolerance of and adaptability to simulated conditions of spaceflight such as confinement, work, monotony, and social/physical isolation that impact behavioral health and performance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 30 and 55 years
* A master's degree (or its equivalency in work experience) in Science, Technology, Engineering and Math (STEM) or military service
* Free of psychological/psychiatric conditions that preclude participation
* BMI < 35
* Ability to read/write English

Exclusion Criteria:

* History of neurological, psychiatric, or other medical condition that excludes participation
* Current mania or psychosis
* Current depression
* Current poor resiliency
* Alcohol or drug abuse in the past year based upon history and urine toxicology screen.
* Current smoker/tobacco user.
* Acute, chronic, or debilitating medical conditions, major Axis I psychiatric illness, epilepsy, or thyroid disease based
* Cardiovascular, neurological, gastrointestinal, or musculoskeletal problems that exclude participation
* For MRI testing any of the following conditions may exclude subjects from participation in the present experiment: Tinnitus; sensorineural hearing loss > 30 decibels; pace maker or internal defibrillator; metallic implants (e.g. orthopedic plates after bone fractures, joint replacements, surgical staples or clips, artificial heart valves, stents, cava filters); metallic splinters (e.g. after an accident or due to war injury); non-removable dental brace; tattoo (some tattoo inks contain metallic particles); permanent make-up; intrauterine contraceptive device; cochlear implant (implanted hearing device); medication pump; acupuncture needle; other foreign bodies/objects which are non-removable; pregnancy (or its possibility); previous brain and/or heart surgery; and fear of tight spaces.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Resilience | Days 1 and 8
  Change in Resilience

SECONDARY OUTCOMES:
Stress | Days 1-8
  Percent change in salivary cortisol
Biomarker-Response to Stress | Days 2, 4, 6, 8
  Percent change in Brain Derived Neurotrophic Factor
Brain Structure | Days 1 and 8
  Change in brain structure using magnetic resonance imaging (MRI)
Brain Function | Days 1 and 8
  Change in brain function using MRI
Cognitive Performance | Days 2-8
  Change in reaction time and accuracy using a computer-based test battery
Sleep Timing and Duration | Days 1-8
  Continuous actigraphy recordings
Heart Rate Monitoring | Days 2, 4, 6, 8
  24 h ECG data will be collected to derive heart rate (HR) and heart rate variability (HRV) measures as a peripheral index of vagal balance.

CONTACTS AND LOCATIONS:
Overall Officials: David Dinges, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No